CLINICAL TRIAL: NCT04416893
Title: Prevalence of SARS -Cov2 Carriage in Asymptomatic and Mildly-symptomatic Children, a Cross-sectional, Prospective, Multicentre, Observational Study in Primary Care-Part 2 After the Lifting of the Lockdown
Brief Title: Part 2 on the Study Prevalence of SARS -Cov2 Carriage in Asymptomatic and Mildly-symptomatic Children (COVILLE2) (WHO)
Acronym: COVILLE2
Status: Withdrawn | Type: Observational
Why Stopped: With the rapid evolution of COVID-19, the objective was no longer relevant
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Association Clinique Thérapeutique Infantile du val de Marne (Other); Groupe de Pathologies Infectieuses Pédiatriques (GPIP) (Other); Francophone Pediatric Resuscitation and Emergency Group (GFRUP) (Other)
Responsible Party: Sponsor
Other Study IDs: COVILLE2
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: COVID19
Keywords: RT-PCR SARS-CoV-2; Serology SARS-CoV-2; Children
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children under 15 years of age in a community: Children under 15 years of age in a community : kindergarten, school, college, holiday center, etc.
  Interventions: Diagnostic Test: RT-PCR SARS-Cov2; Diagnostic Test: Sars-Cov2 serology

INTERVENTIONS:
Diagnostic Test: RT-PCR SARS-Cov2 — nasopharyngeal swab will be taken for detection of SARS-CoV-2 by RT-PCR
Diagnostic Test: Sars-Cov2 serology — A microsample of blood will be taken for serology

SUMMARY:
France and in particular the paris area was one of the countries most affected by the pandemic Covid19.

School closures and a generalized lockdown of the population were instituted in France from 17 March 2020 to 10 May 2020. Schools and nurseries have reopened partially since 11 May 2020. From 2 June, this reopening is more widespread. By combining the search for SARS-Cov2 viruses by PCR and micro-method serology we will be able to evaluate both the infection at a given time and also older contact with SARS-CoV2.

The temporal knowledge of the prevalence of SARS-Cov2 carriage and the serological status (IgM and IgG) after return to the community are crucial information to evaluate the speed of spread of the virus in children. This is the objective of COVILLE2, phase 2 of the COVILLE study.

ELIGIBILITY:
Inclusion Criteria:

* Birth to 15 years old
* taking over the community (kindergarten, school, college, holiday centre, etc.) for at least 1 week

Exclusion Criteria:

* refusal to participate

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children under 15 years of age in a community (kindergarten, school, college, holiday centre, etc.).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of asymptomatic children or children with mild respiratory symptoms | At inclusion
  Proportion of asymptomatic children or children with mild respiratory symptoms (mildly-symptomatic children) with a positive SARS-Cov2 Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) on rhino pharyngeal swab or/and IgM/IgG positive serology in Paris area

SECONDARY OUTCOMES:
Cov2-SARS cases by age | At inclusion
Cov2-SARS cases by symptoms | At inclusion
Viral load | At inclusion
  The viral load of children with SARS-Cov2 positive Reverse Transcriptase Polymerase Chain Reaction depending on the symptoms and the age of the patients
Presence of anti-SARS-CoV-2 antibodies (IgM and IgG) by the rapid serological test | At inclusion

IPD SHARING:
Plan to Share IPD: No